CLINICAL TRIAL: NCT02151032
Title: Using Multimedia Approaches to Communicate Probabilities in Patient Decision Aids for Low-Literacy Populations: Randomized Trial
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Foundation for Informed Medical Decision Making (Other)
Responsible Party: Sponsor
Other Study IDs: 2011-0632; 0619-1 (Other Grant/Funding Number: Foundation for Informed Medical Decision Making)
Record Dates: First submitted 2014-05-27; First posted 2014-05-30 (Estimated); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer; Colorectal cancer screening; Multimedia; Booklet; Pamphlet; Audio CD; Video with animated images; Video with non-moving images; Questionnaires; Surveys
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Videotape Recording; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Colorectal Cancer Screening Booklet + Audio CD: Participants read the booklet about colorectal cancer screening tests, and listen to an audio CD that will narrate the booklet. Questionnaire completion before and after viewing the program.
  Interventions: Behavioral: Booklet; Behavioral: Audio CD; Behavioral: Questionnaires
- Video with Non-Moving Images on iPad: Participants watch a video with non-moving images about colorectal cancer screening tests on an iPad. Questionnaire completion before and after viewing the program.
  Interventions: Behavioral: Video with Non-Moving Images; Behavioral: Questionnaires
- Video with Animated Images on iPad: Participants watch a video with animated images about colorectal cancer screening tests on an iPad. Questionnaire completion before and after viewing the program.
  Interventions: Behavioral: Video with Animated Images; Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Booklet — Participants read a booklet about colorectal cancer screening tests.
  Other Names: Pamphlet
  Groups: Colorectal Cancer Screening Booklet + Audio CD
Behavioral: Audio CD — Participants listen to an audio CD that will narrate the colorectal cancer screening tests booklet.
  Groups: Colorectal Cancer Screening Booklet + Audio CD
Behavioral: Video with Non-Moving Images — Participants watch a video with non-moving images about colorectal cancer screening tests on an iPad.
  Groups: Video with Non-Moving Images on iPad
Behavioral: Video with Animated Images — Participants watch a video with animated images about colorectal cancer screening tests on an iPad.
  Groups: Video with Animated Images on iPad
Behavioral: Questionnaires — Questionnaire completion before and after viewing the program.
  Other Names: Surveys

SUMMARY:
The goal of this research study is to compare how people who are 45-75 years old respond to 3 different versions of a program about screening tests for colorectal cancer. Researchers want to use this study as part of a long-term project to learn the best ways to communicate health information to patients.

DETAILED DESCRIPTION:
If you agree to take part in this study, you will be randomly assigned (as in a roll of dice) to 1 of 3 study groups. Neither you nor the study staff will be able to choose which group you will be in:

* If you are in Group 1, you will read a booklet about colorectal cancer screening tests. While reading the booklet, you will also listen to an audio CD that will narrate the booklet.
* If you are in Group 2, you will watch a video with non-moving images about colorectal cancer screening tests on an iPad.
* If you are in Group 3, you will watch a video with animated images about colorectal cancer screening tests on an iPad.

You will complete questionnaires before and after viewing the program that will contain questions about:

* Your age and what language you speak
* Your math and reading comprehension
* Your knowledge of colorectal cancer and colorectal cancer screening
* Your thoughts about colorectal cancer screening
* Your opinions about this study, and
* How well you understand the booklet/video you view as part of this study

It will take about 1 hour to complete all the questionnaires. In total, the study will take about 1 ½ to 2 hours to complete. After you have completed the questionnaires, your participation in the study will be over.

This is an investigational study.

Up to 201 people will take part in this multicenter study. Up to 67 will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women 45 to 75 years of age.
2. Participant must speak English.

Exclusion Criteria:

1) Self-reported diagnosis of colon cancer.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants from MD Anderson Cancer Prevention Center (CPC), Literacy Advance of Houston (LAH), Ephiphany Community Health Outreach Services (ECHOS), and Bethel's Heavenly Hands
Sampling Method: Probability Sample
Enrollment: 189 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2020-05-19 (Actual); Study Completion 2020-05-19 (Actual)

PRIMARY OUTCOMES:
Gist and Verbatim Knowledge for a Colorectal Cancer Screening Program | 1 day
  The fixed effects analysis of variance (ANOVA) will utilize a factorial design with two factors: content presentation type (standard, animated, interactive) and numeracy status (high and low based on US population scores). Main dependent measures are gist and verbatim knowledge. Gist and verbatim knowledge scores (0-100) looked at separately as well as combined.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Volk, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (4):
- United States (4):
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Bethel's Heavenly Hands, Houston, Texas
  - Literacy Advance of Houston, Houston, Texas
  - Ephiphany Community Health Outreach Services, Houston, Texas

REFERENCES:
- [Derived] Housten AJ, Kamath GR, Bevers TB, Cantor SB, Dixon N, Hite A, Kallen MA, Leal VB, Li L, Volk RJ. Does Animation Improve Comprehension of Risk Information in Patients with Low Health Literacy? A Randomized Trial. Med Decis Making. 2020 Jan;40(1):17-28. doi: 10.1177/0272989X19890296. Epub 2019 Dec 3. PMID 31795820
- [Derived] Housten AJ, Lowenstein LM, Hoover DS, Leal VB, Kamath GR, Volk RJ. Limitations of the S-TOFHLA in measuring poor numeracy: a cross-sectional study. BMC Public Health. 2018 Mar 27;18(1):405. doi: 10.1186/s12889-018-5333-9. PMID 29587709
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org